CLINICAL TRIAL: NCT02926443
Title: Effectiveness of the Upper Extremity Neuromuscular Training Program (UpEx-NTP) on Shoulder Function of People With Rotator Cuff Tendinopathies: A Pilot Randomized Control Trial
Brief Title: Effectiveness of Supervised Motor Control Exercises on Rotator Cuff Tendinopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: CIRRIS (Center for Interdisciplinary Research in Rehabilitation and Social Integration) (Unknown); OPPQ (Ordre Professionnel de la Physiothérapie du Québec) (Unknown); REPAR (Réseau Provincial de Recherche en Adaptation-Réadaptation) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-446
Record Dates: First submitted 2016-07-18; First posted 2016-10-06 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Shoulder Impingement Syndrome; Shoulder Rotator Cuff Tendinopathy
Keywords: Shoulder; Motor control; Usual physiotherapy care; Supervised exercise program
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One-on-one Usual Physiotherapy Care (Control) (Active Comparator): The Ctl group (n =16) will receive physiotherapy usual care treatments during a 6-week period. The Ctl group will receive 2 physiotherapy treatments (30 minutes) in the clinic per week (total of 12 treatments) as well as an individualized home exercise program (HEP). Treatments will include range of motion exercises, manual therapy treatments, modalities, and strengthening exercises, as determined by the treating physiotherapist. Specific muscle group exercises and parameters will be documented by the treating physiotherapist on a provided summary sheet.
  Interventions: Other: Usual Physiotherapy Care
- Group Program (UpEx-NTP) (Exp) (Experimental): The Exp group (n =16) will partake in a 6-week group Upper Extremity Neuromuscular Training Program that consists of postural education, strength exercises, motor control exercises, and upper extremity functional tasks common for active military personnel. The UpEx-NTP program consists of 35-45 minutes of exercise, three times a week for 6 weeks (18 treatments), supervised by a physiotherapist. The program consists of 11 stations with several variations of difficulty of the same exercise per station. The exercises of each station will be performed in order of difficulty. The participant chooses one exercise to perform per station based on their current ability while respecting their pain levels at 3/10 or less.
  Interventions: Other: Upper Extremity Neuromuscular Training Program

INTERVENTIONS:
Other: Upper Extremity Neuromuscular Training Program — Neuromuscular and strengthening shoulder exercises in a group setting.
  Arms: Group Program (UpEx-NTP) (Exp)
Other: Usual Physiotherapy Care — One-on-one physiotherapy care in a clinical setting.
  Arms: One-on-one Usual Physiotherapy Care (Control)

SUMMARY:
The shoulder is the most mobile joint in the body but still has the responsibility of ensuring a strong stability of our upper limbs during daily activities. The shoulder joint therefore requires a significant level of neuromuscular control at all times. The shoulder heavily relies on 4 key stabilizing muscles, known as the rotator cuff complex (RC). A tendinopathy of the RC may cause pain, significant muscle weakness, and a decrease in motor control of the shoulder during functional activities as well as work tasks. Individuals who have an RC tendinopathy often have neuromuscular and proprioceptive deficits. The objectives of this study are to evaluate the effectiveness of a brand new group strength and motor control exercise program for the upper extremities and to compare the effectiveness of this program to usual one-on-one physiotherapy care (such as manual therapy, motion exercises, strengthening, manual techniques) in reducing shoulder pain and improving overall function. A total of 33 participants suffering from an RC tendinopathy have been recruited; 16 have been assigned to the exercise group (EXP) and 17 participants have received usual physiotherapy care (CTL). Participants in the EXP group partook in the new exercise program 3 times / week for 6 weeks whereas participants in the CTL group received usual physiotherapy treatments twice / week with home exercises for 6 weeks. The results of this study will provide clinicians with a cost-effective and innovative treatment approach to treating shoulder pain. This study will provide active rehabilitation guidelines for reducing shoulder pain and the incidence of recurrence.

DETAILED DESCRIPTION:
The importance of our shoulders to everyday movement and activity is often not fully appreciated, until we are limited by injury or pain. The shoulder complex allow us to interact with our surroundings while acting as the functional link between our stable trunks and our free moving upper limbs. This is no easy task for highly mobile joints such as the shoulders. A shoulder injury can be functionally devastating to an individual, and can potentially place unnecessary financial stress on our health care system. Shoulder pain is currently among the most common reasons to visit a general practitioner or a physiotherapist today. Shoulder pain is third in prevalence, only to back and neck pain, and nearly two-thirds of adults suffer from shoulder pain at some point during their lives. Despite being an important focus for rehabilitative care, we have yet to confidently establish efficient and potentially cost effective methods for treating shoulder pathologies and pain. Among shoulder disorders, the rotator cuff (RC) muscles are the leading source of shoulder pain. Due to the vast mobility of the shoulder complex, it relies greatly on the stability and control provided by its supportive tissues, notably the rotator cuff muscles; often rendering them highly susceptible to injury. It has been noted that individuals affected by rotator cuff tendinopathies (RCt) often exhibit motor control and shoulder proprioception deficits. As noted by Cools and colleagues, rehabilitative training programs that focus on motor control are greatly needed for rehabilitation as well as to prevent re-injury. Accordingly, rehabilitation interventions should focus on motor (re)learning, targeting a better muscle coordination to reduce motor control impairments, optimize movement control, and improve muscle strength.

Motor control rehabilitation: To address the motor control deficits among individuals affected by an RCt, we have developed a novel, structured, and supervised group exercise-based program focusing on neuromuscular reeducation. It is well documented in the scientific literature that motor control and proprioception exercises are crucial for healing among this population. However, the effectiveness of a group delivery method remains unknown. It is presently unclear how a group exercise program compares to one-on-one physiotherapy care for shoulder dysfunctions. The developed group program allows patients to individually progress their exercises based on their symptoms, while being guided and corrected by the supervising physiotherapist. This model allows several patients to access physiotherapy services simultaneously, while remaining cost and resource effective for the clinics. To appreciate the goal of the proposed exercise program, it is important to understand the physiological and biomechanical factors directly related to shoulder stability.

Underlying mechanisms for shoulder stability: For its joint stability, the glenohumeral (GH) joint heavily depends on muscle strength, adequate synergistic activity between the neuromuscular structures, as well as a strong joint position sense (a subcategory of proprioception). Our ability to detect our limbs in space helps us to interact with our surroundings and contributes to the neuromuscular stability of our joints. A RCt is often associated with a subacromial impingement syndrome, where structures under the acromion become pinched during arm elevation. Such a compression during arm movements can include abnormal shoulder kinematics, as well as RC and scapular muscles performance deficits. This inadequate scapulothoracic muscle control is believed to contribute to a reduction of amplitude in posterior tilting and lateral rotation of the scapula, which causes the acromion to remain in a lower anterolateral position resulting in a dynamic narrowing of the subacromial space. Also, the abnormal muscle control is associated with superior migration of humeral head with respect to the glenoid fossa, which again leads to a dynamic narrowing of the subacromial space. These deficits contribute to the impingement of subacromial structures and often lead to the symptoms associated with an RCt. What makes the investigated approach unique in addressing RC disorders is the resource-effective exercise rehabilitation model the investigators propose; a motor control and strengthening approach well supported in the scientific literature and packaged in a conveniently resource-friendly protocol. This approach maximizes patient autonomy while being matched to a suitable level of physiotherapist supervision. The investigators believe that the Upper Extremity Neuromuscular Training Program (UpEx-NTP) provides a realistic and financially beneficial solution to a costly health care problem.

Research Question: How will a 6-week UpEx-NTP improve shoulder function, pain, and joint position sense (JPS) in individuals affected by a rotator cuff (RC) tendinopathy compared to usual physiotherapy care? The primary objective of this randomized control trial (RTC) is to compare, in terms of symptoms and functional limitations, a group receiving a group-supervised rehabilitation program (UpEx-NTP) centered on strength and motor control training to a group receiving usual one-on-one physiotherapy clinical care in individuals affected by a RC tendinopathy of the shoulder. It is hypothesized that both the UpEx-NTP (Exp) and usual physiotherapy care (Ctl) groups will equally demonstrate statistically (p-value < 0.05) and clinically (all noted changes above their MCID : DASH questionnaire = 11 points, WORC index = 12 points and the Numeric Rating Scale for pain = 2 points) significant changes in shoulder function and pain over a 6-week period in individuals with an RC tendinopathy and will be maintained over time, notably 12-weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Reported pain and / or stiffness to shoulder joint, localized tenderness over one of the rotator cuff muscles, reported night pain to the shoulder,
2. Painful arc of movement during flexion or abduction,
3. Positive Neer's Test or Kennedy-Hawkins Test,
4. Pain on resisted external (lateral) rotation, abduction or Empty Can Test,
5. A combined DASH-CF (Disability of the Arm, Shoulder, and Hand - Canadian French) score (all 3 subsections) greater than 15%, or a WORC-CF (Western Ontario Rotator Cuff Index - Canadian French) score greater than 12%,
6. Active military members.

N.B. The minimal scores for both the DASH and WORC questionnaires are based on their minimal clinically important difference (MCID). Also, the combination of criteria 2), 3) and 4) have a good diagnostic accuracy with sensitivity and specificity values ≥ 0.74. and Positive Likelihood Ratio = 3.5.

Exclusion Criteria:

1. Any prior history of shoulder surgery, dislocations, fractures, capsulitis,
2. Demonstrate any systematic pathologies (such as diabetes, neurological signs or symptoms, complex regional pain syndrome, rheumatoid conditions, or signs and symptoms of vascular compression or vestibular dysfunction),
3. Not able to commit to the treatment schedule of the project.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-01; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in self-reported shoulder function at 6 weeks (DASH-CF) | Baseline to 6 weeks
  DASH-CF: Disability of Arm, Shoulder, and Hand Questionnaire (Canadian French). Self-reporting questionnaire that assesses the upper limb pain and disability of the participants. The DASH has 30-items over three sub-sections: General, Work, and Sports / Art. You can also interpret the global score (sum of the 3 sections). The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability)-this is called the DASH score.

SECONDARY OUTCOMES:
Change from baseline in self-reported shoulder function specific to rotator cuff disorders at 6 months (WORC-CF) | Baseline to 6 weeks
  WORC-CF: Western Ontario Rotator Cuff Index Questionnaire (Canadian French). A self-reporting, disease-specific quality of life questionnaire, that will evaluate the change in symptoms of our participants specific to their rotator cuff disorder.
Change from baseline in self-reported shoulder function specific to rotator cuff disorders at 6 weeks (WORC-CF) | Baseline to 12 weeks
  WORC-CF: Western Ontario Rotator Cuff Index Questionnaire (Canadian French). A self-reporting, disease-specific quality of life questionnaire, that will evaluate the change in symptoms of our participants specific to their rotator cuff disorder.
Change from baseline in shoulder strength at 6 weeks | Baseline to 6 weeks
  Bilateral shoulder strength will be assessed using a hand held dynamometer (HHD) by the evaluator for shoulder abductors and external rotator muscles.
Change from baseline in level of perceived shoulder pain at 6 weeks (NPRS) | Baseline to 6 weeks
  Pain levels will be assessed at 6 weeks using the 11-point Numeric Rating Scale (NRS) for pain, where 0 represents "no pain" and 10 represents "worst pain imaginable".
Change from baseline in common military task | Baseline to 6 weeks
  Repeated sand bag lift (20kg, 30 repetitions in 3 minutes 30 seconds)
Change from baseline of perceived level of change in symptoms | Baseline to 6 weeks
  Global Rating of Change (GROC) questionnaire
Change from baseline of perceived level of change in symptoms | Baseline to 12 weeks
  Global Rating of Change (GROC) questionnaire
Change from baseline in self-reported shoulder function at 12 weeks (DASH-CF) | Baseline to 12 weeks
  DASH-CF: Disability of Arm, Shoulder, and Hand Questionnaire (Canadian French). Self-reporting questionnaire that assesses the upper limb pain and disability of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Luc J. Hébert, MSc PT, PhD, Study Director — CIRRIS / IRDPQ, Canadian Armed Forces (CAF); Jean-Sébastien Roy, MSc PT, PhD, Study Director — IRDPQ and CIRRIS
Locations (1):
- Valcartier Garrison, Physiotherapy Clinic, Shannon, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ager AL, Roy JS, Gamache F, Hebert LJ. The Effectiveness of an Upper Extremity Neuromuscular Training Program on the Shoulder Function of Military Members With a Rotator Cuff Tendinopathy: A Pilot Randomized Controlled Trial. Mil Med. 2019 May 1;184(5-6):e385-e393. doi: 10.1093/milmed/usy294. PMID 30423137